CLINICAL TRIAL: NCT00288236
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind, Parallel-Group, Fixed-Dose Study Evaluating the Effect of One Dose of Rimonabant (20 mg/Day) on Glycemic Control in Type 2 Diabetic Patients Inadequately Controlled With Insulin
Brief Title: Study Evaluating Rimonabant Efficacy in Insulin-Treated Diabetic Patients(ARPEGGIO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC5593
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Rimonabant (SR141716)
Drug: Placebo

SUMMARY:
Primary: Effect on HbA1c over 48 weeks in insulin-treated patients with type 2 diabetes

Secondary: Effect on glucose, total daily insulin dose, body weight, waist circumference, HDL-cholesterol, triglycerides - Safety, tolerability

DETAILED DESCRIPTION:
The total duration of the study will be up to 360 days including screening period (up to 14 days) and double-blind treatment period (approximately 11 months).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged greater than or equal to 18 years.
* Diagnosis of type 2 diabetes as defined by WHO criteria.
* Type 2 diabetes treated with insulin for at least 3 months (insulin dose of at least 30 U/day for at least 4 weeks).
* HbA1C greater than or equal to 7%.
* Having signed the informed consent form.

Exclusion Criteria:

General:

* Weight loss > 5 kg within 3 months prior to screening visit.
* Pregnancy or lactation.
* Absence of medically approved contraceptive methods for females of childbearing potential.
* Administration of other investigational drugs within 30 days prior to screening visit.
* Previous participation in a Rimonabant study.
* Presence or history of allergic reaction or intolerance to multiple drugs.

Related to endocrine and metabolic disorders:

* Presence of any clinically significant endocrine disease according to the Investigator.Note: euthyroid patients on replacement therapy will be included if the dosage of thyroxine is stable for at least 3 months prior to screening visit.
* Fasting C-peptide < 1.0 ng/mL.

Related to other disorders:

* Presence of any severe medical or psychological condition that in the opinion of the Investigator would compromise the patient's safety or successful participation in the study.
* Presence or history of cancer within the past 5 years with the exception of adequately treated localized basal cell skin cancer or in situ uterine cervical cancer.

Related to laboratory findings:

* Positive test for hepatitis B surface antigen and/or hepatitis C antibody.
* Abnormal TSH level (TSH > ULN or < LLN).
* Positive urine pregnancy test.

Related to previous or concomitant medications:

* Antidiabetic drugs other than insulin within 3 months prior to screening visit.
* Drugs affecting weight (e.g., sibutramine, orlistat, herbal preparations, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2006-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Absolute change in HbA1C from baseline to Week 48

SECONDARY OUTCOMES:
Fasting glucose, total daily insulin dose, body weight, waist circumference, HDL-cholesterol, triglycerides, safety (physical examination, vital signs, laboratory tests, adverse events).

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (12):
- Sanofi-Aventis, Bridgewater, New Jersey, United States
- Sanofi-Aventis, Buenos Aires, Argentina
- Sanofi-Aventis, Lane Cove, Australia
- Sanofi-Aventis, Laval, Canada
- Sanofi-Aventis, Providencia, Chile
- Sanofi-Aventis, Paris, France
- Sanofi-Aventis, Berlin, Germany
- Sanofi-Aventis, Milan, Italy
- Sanofi-Aventis, Gouda, Netherlands
- Sanofi-Aventis, Moscow, Russia
- Sanofi-Aventis, Midrand, South Africa
- Sanofi-Aventis, Guildford, United Kingdom